CLINICAL TRIAL: NCT02052765
Title: AnalyST & Brugada Syndrome - Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR-10-022-FR-HV
Record Dates: First submitted 2011-09-19; First posted 2014-02-03 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ajmaline test (Experimental): All patients underwent ajmaline test for ST shift recording
  Interventions: Device: ECG continuous recording (Analyze ST)

INTERVENTIONS:
Device: ECG continuous recording (Analyze ST) — During the ajmaline test, continuous ECG recording was forced to record ST shift
  Other Names: Analyze ST

SUMMARY:
Brugada syndrome is characterized by a ST shift on the surface ECG, and a specific morphology of the Twave. This ECG abnormality is called a type 1-ECG, and is variable in time. Patients presenting a Brugada syndrome are exposed to sudden cardiac death, although it's difficult to predict patients at high risk. It is suspected that the type 1-ECG burden might be correlated to the ventricular fibrillation risk of these patients, but there is no mean to record the ECG over a long period of time.

The objective of the study is to evaluate the correlation between ST elevation on the electrocardiogram (ECG) and ST shift on the intracardiac electrograms (EGM) recorded with the AnalyST ICD, to assess the ability of the device to detect the type 1-ECG. Patients enrolled in the study are patients already implanted with a defibrillator for their Brugada syndrome. During an Ajmalin test, which unmasks the type 1-ECG, both intracardiac EGM and surface ECG will be compared to assess the detection of the typical ST-shift by the ICD.

DETAILED DESCRIPTION:
To evaluate the correlation between ST elevation on the ECG and ST shift on the intracardiac EGM recorded with the AnalyST ICD, patients enrolled will have to be already diagnosed as presenting the Brugada Syndrome. They will undergo an ajmaline test, to unmask the type 1-ECG, characteristic from the Brugada syndrome.During the test, both surface ECG and intracardiac signal will be continuously recorded; then the signals will be compared in terms of amplitude of the ST shift, duration of the shift, and recovery period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Brugada syndrome and previous positive Ajmalin test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
ST shift correlation | Acute testing - 4h after the beginning of the ajmaline test.
  Correlation between external ECG - ST elevation and device-recorded ST shift. The ajmaline is the reference method to unmask type 1-ECG in Brugada syndrome. During an ajmaline test, both surface ECG and intracardial EGM will be continuously recorded and compared to allow comparison of the signals in terms of amplitude and duration of the ST shift and recovery timing.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Probst, M.D., Principal Investigator — Hopital Laennec
Locations (1):
- Hopital Laennec, Nantes, France